CLINICAL TRIAL: NCT01195844
Title: Rotavirus Gastroenteritis in Children Up to 5 Years of Age. Surveillance Performed in Hospitals From Four Brazilian Regions.
Brief Title: Gastroenteritis From Rotavirus Infection in Brazilian Children Less Than 5 Years of Age (Study V260-031).
Status: Terminated | Type: Observational
Why Stopped: Inadequate recruitment
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: V260-031
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Results first posted 2012-12-05 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-02

CONDITIONS: Pediatric Gastroenteritis
Keywords: Pediatric gastroenteritis, rotavirus infection
MeSH Terms: conditions — Rotavirus Infections | interventions — Rotavirus Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Brazilian Children With Rotavirus Gastroenteritis: Brazilian children under 5 years of age who have diarrhea attributed to rotavirus located in 4 hospitals from 4 different Brazilian regions
  Interventions: Biological: Rotavirus Vaccine

INTERVENTIONS:
Biological: Rotavirus Vaccine — This is an observational study evaluating hospitalizations and the medical care for the treatment of diarrhea from rotavirus infection in children < 5 years of age; however, any rotavirus vaccines used in the children presenting with rotavirus-attributed diarrhea were evaluated, as well the prevalent rotavirus serotypes in this sample for future vaccine development.

SUMMARY:
This is a 1-year study evaluating hospitalizations and the medical care for the treatment of diarrhea from rotavirus infection in children < 5 years of age, conducted in four hospitals located in four Brazilian regions. A stool sample from each eligible child passing 3 or more loose stools or watery stools within a period of 24 hours and requiring hospitalization or rehydration therapy (oral or IV rehydration) will be tested for the presence of rotavirus, using standard laboratory procedures (ie, Enzyme Linked Ligand Sorbent Assay, or ELlSA) by all participating hospitals.

ELIGIBILITY:
Inclusion Criteria:

* a child < 5 years of age being treated for acute gastroenteritis within 72 hours prior to evaluation in the study hospitals.
* outpatient children < 5 years of age submitted for treatment of acute gastroenteritis within 72 hours prior to evaluation in the study clinics.

Exclusion Criteria:

* none specified

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children less than 5 years of age from four Brazilian cities with diarrhea attributed to rotavirus infection.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2010-08; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Divina das Dores P Cardoso, Doctor, Principal Investigator — Instituto de Patologia Tropical e Saúde Pública IPTSP-UFG; Edson Moreira, MD, PhD, Principal Investigator — Hospital Santo Antonio - Obras Sociais Irma Dulce; Alfredo Gilio, MD, Principal Investigator — Hospital Universitário da Universidade de Sao Paulo; Paulo Carvalho, MD, Principal Investigator — Hospital de Clínicas da Universidade Federal do Rio de Grande do Sul

RESULTS

PARTICIPANT FLOW:
Groups:
- Children Hospitalized For Diarrhea: Children up to 5 years of age hospitalized for diarrhea in the 4 Brazilian hospital research centers
Period: Overall Study
Arm/Group | Children Hospitalized For Diarrhea
Started | 230
Completed | 190
Not Completed | 40
Not completed — Fecal sample not collected | 40

BASELINE CHARACTERISTICS:
Groups:
- Children Who Provided a Fecal Sample: Children up to 5 years of age hospitalized for diarrhea and providing a fecal sample in the 4 Brazilian hospital research centers. Diarrhea was defined as the passage of 3 or more soft/liquid feces in a 24-hour period.
Arm/Group | Children Who Provided a Fecal Sample
Number analyzed (Participants) | 190
Age, Customized [Number; unit: participants] | 190
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84
  Male | 106
Rotavirus Vaccination Received [Number; unit: Participants]
  Yes | 175
  No | 15

OUTCOME MEASURES:

1. Primary Outcome: The Number of Hospitalizations for Diarrhea in Children up to 5 Years of Age
Description: The total number of hospitalizations for diarrhea in children up to 5 years of age in the 4 Brazilian hospital research centers was reported. Diarrhea was defined as the passage of 3 or more soft/liquid feces in a 24-hour period.
Time Frame: 1 year
Population: The population analyzed was all enrolled participants whether or not a fecal sample was obtained
Measure: Number; unit: participants
Groups:
- Children Hospitalized For Diarrhea: Children hospitalized for diarrhea in the 4 Brazilian hospital research centers
Arm/Group | Children Hospitalized For Diarrhea
Number analyzed (Participants) | 230
participants | 230

2. Primary Outcome: The Percentage of Hospitalizations for Diarrhea in Children up to 5 Years of Age
Description: The percentage of total hospitalizations for children up to 5 years of age in the 4 Brazilian hospital research centers that were for diarrhea. Diarrhea was defined as the passage of 3 or more soft/liquid feces in a 24-hour period.
Time Frame: 1 year
Population: The population to be analyzed was all hospitalizations for any reason for children up to 5 years of age in the 4 hospital research centers
  The number of total hospitalizations for children up to 5 years of age was not known; thus this outcome measure was not evaluated
Arm/Group | Children Hospitalized for Diarrhea
Number analyzed (Participants) | 0

3. Primary Outcome: The Geographic Distribution of Hospitalizations for Diarrhea That Are Caused by Rotavirus
Description: Children up to 5 years of age hospitalized for diarrhea were tested for fecal rotavirus as determined by enzyme immunoassay. Diarrhea was defined as the passage of 3 or more soft/liquid feces in a 24-hour period. For each geographic location, the number of hospitalizations for diarrhea that was caused by rotavirus was reported.
Time Frame: 1 year
Population: The population analyzed was children up to 5 years of age hospitalized for diarrhea. A total of 190 of the 230 participants had fecal samples analyzed; 27 of these had stool samples positive for rotavirus.
Measure: Number; unit: Participants
Groups:
- Salvador (Northeast): Children up to 5 years of age hospitalized for diarrhea that tested positive for rotavirus in the Salvador (Northeast Brazil) hospital research center
- Goiânia (Center-West): Children up to 5 years of age hospitalized for diarrhea that tested positive for rotavirus in the Goiânia (Center-West Brazil) hospital research center
- Porto Alegre (South): Children up to 5 years of age hospitalized for diarrhea that tested positive for rotavirus in the Porto Alegre (South Brazil) hospital research center
- São Paulo (Southeast): Children up to 5 years of age hospitalized for diarrhea that tested positive for rotavirus in the São Paulo (Southeast Brazil) hospital research center
Arm/Group | Salvador (Northeast) | Goiânia (Center-West) | Porto Alegre (South) | São Paulo (Southeast)
Number analyzed (Participants) | 55 | 101 | 8 | 26
Participants | 17 | 3 | 0 | 7

4. Primary Outcome: The Percentage of Hospitalizations for Diarrhea That Are Caused by Rotavirus
Description: Children up to 5 years of age hospitalized for diarrhea were tested for fecal rotavirus as determined by enzyme immunoassay. Diarrhea was defined as the passage of 3 or more soft/liquid feces in a 24-hour period. The number of hospitalizations for diarrhea from rotavirus infection was divided by the total number of hospitalizations for diarrhea in the 4 hospital research centers.
Time Frame: 1 year
Population: Children hospitalized for diarrhea and providing a fecal sample in the 4 Brazilian hospital research centers
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Children Hospitalized For Diarrhea Who Provided a Fecal Sample: Children up to 5 years of age hospitalized for diarrhea and providing a fecal sample in the 4 Brazilian hospital research centers
Arm/Group | Children Hospitalized For Diarrhea Who Provided a Fecal Sample
Number analyzed (Participants) | 190
percentage of participants | 14.2 [12.49 to 15.93]

5. Primary Outcome: The Number of Hospitalizations for Diarrhea That Are Caused by Rotavirus by Age Group
Description: Children up to 5 years of age hospitalized for diarrhea were tested for fecal rotavirus as determined by enzyme immunoassay. Diarrhea was defined as the passage of 3 or more soft/liquid feces in a 24-hour period. The number of hospitalizations for diarrhea from rotavirus infection was reported for each age group.
Time Frame: 1 year
Population: The population analyzed was the 27 of 190 participants who had a fecal sample positive for rotavirus.
Measure: Number; unit: participants
Groups:
- Children Hospitalized For Rotavirus-Positive Diarrhea: Children up to 5 years of age hospitalized for diarrhea that tested positive for rotavirus in the 4 Brazilian hospital research centers
Arm/Group | Children Hospitalized For Rotavirus-Positive Diarrhea
Number analyzed (Participants) | 27
participants
  Age 0 to 3 months | 2
  Age 4 to 6 months | 0
  Age 7 to 9 months | 0
  Age 10 to 12 months | 1
  Age 13 to 15 months | 3
  Age 16 to 18 months | 2
  Age 19 to 21 months | 1
  Age 22 ato 24 months | 3
  Age 25 to 36 months | 8
  Age 37 to 48 months | 3
  Age >48 months | 4

6. Primary Outcome: The Numbers of Participants Hospitalized for Diarrhea and Rotavirus-caused Diarrhea Per Month
Description: Children up to 5 years of age hospitalized for diarrhea were tested for fecal rotavirus as determined by enzyme immunoassay. Diarrhea was defined as the passage of 3 or more soft/liquid feces in a 24-hour period.
Time Frame: 1 year
Population: The population analyzed was all enrolled participants whether or not a fecal sample was obtained
Measure: Number; unit: Participants
Groups:
- Total Number Hospitalized For Diarrhea of Any Cause: Total number of children up to 5 years of age hospitalized for diarrhea of any cause in the 4 Brazilian hospital research centers
- Total Number Diagnosed With Rotavirus Diarrhea: Children up to 5 years of age diagnosed with rotavirus diarrhea in the 4 Brazilian hospital research centers
Arm/Group | Total Number Hospitalized For Diarrhea of Any Cause | Total Number Diagnosed With Rotavirus Diarrhea
Number analyzed (Participants) | 230 | 27
Participants
  January 2010 | 1 | 0
  August 2010 | 41 | 5
  September 2010 | 24 | 8
  October 2010 | 7 | 2
  November 2010 | 23 | 0
  December 2010 | 7 | 0
  January 2011 | 5 | 0
  February 2011 | 14 | 1
  March 2011 | 6 | 0
  April 2011 | 12 | 2
  May 2011 | 18 | 0
  June 2011 | 16 | 2
  July 2011 | 22 | 2
  August 2011 | 18 | 4
  September 2011 | 13 | 1
  October 2011 | 2 | 0
  November 2011 | 1 | 0

7. Primary Outcome: The Duration of Hospitalization for Participants Enrolled in the Study
Description: The mean duration (days) of hospital stay for children up to 5 years of age hospitalized for diarrhea in the 4 Brazilian hospital research centers. Diarrhea was defined as the passage of 3 or more soft/liquid feces in a 24-hour period.
Time Frame: From hospital admission to discharge
Population: The population analyzed was all enrolled participants whether or not a fecal sample was obtained.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Children Hospitalized For Diarrhea
Number analyzed (Participants) | 230
days | 1.83 (2.65)

8. Primary Outcome: The Number of Deaths in Hospitalized Participants Enrolled in the Study
Description: The number of deaths among children up to 5 years of age hospitalized for diarrhea in the 4 Brazilian hospital research centers. Diarrhea was defined as the passage of 3 or more soft/liquid feces in a 24-hour period.
Time Frame: 1 year
Population: Participants were not followed-up in the study; thus the number of deaths was not known.
Arm/Group | Children Hospitalized For Diarrhea
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events were not collected in this observational study
Arm/Group | Children Hospitalized For Diarrhea
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The initial publication of this study will be multicenter, comprising data from all sites involved. After the multicenter publication, or 24 months after the end of the study, each site involved may publish its own results in an independent fashion.

The sponsor will also have the opportunity to review all the proposed abstracts,

manuscripts or lectures related to this study 60 days before submission for

publication/presentation.